CLINICAL TRIAL: NCT05981469
Title: Can Cervical Stiffness Predict Successful Vaginal Delivery After Induction of Labour?
Acronym: CASPAR
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool Women's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UoL001713
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Induced Vaginal Delivery
Keywords: cervical stiffness; induction of labour

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Induction of labour
  Interventions: Device: Cervical Stiffness Assessmenr; Other: Bishop's Score Assessment

INTERVENTIONS:
Device: Cervical Stiffness Assessmenr — The cervical stiffness is assessed by using the licensed, CE-marked Pregnolia System, during a sterile speculum examination. The single-use, sterile Pregnolia Probe is placed on the anterior lip of the cervix at 12 o'clock position and a recording of cervical stiffness is generated over maximum 60 seconds (typically ̴15 seconds) and displayed as Cervical Stiffness Index (CSI) in mbar. The measurement is repeated 3 consecutive times without any time lag.
Other: Bishop's Score Assessment — Sterile digital vaginal examination to illicit the Bishop's score (0-12).

SUMMARY:
The purpose of this study is to determine if a new antenatal test of cervical stiffness can be used to predict which patients will have a successful vaginal delivery following an induction of labour.

A licensed, CE-marked, vacuum-aspiration device called the Pregnolia system has been developed to give quantitative cervical stiffness index score during pregnancy. The CASPAR study will compare cervical stiffness scores to bishop's scores prior to induction of labour and correlate the results to the outcome of delivery.

DETAILED DESCRIPTION:
CASPAR is a single site prospective, exploratory, cohort study of 100 women with singleton pregnancy undergoing induction of labour at the Liverpool Women's Hospital (LWH).

All eligible participants giving written informed consent will be asked to undergo a sterile speculum examination for cervical stiffness assessment, prior to routine vaginal digital examination for Bishop's score assessment. Participants will then proceed with their induction of labour as per the unit policy.

Once recruited the participants will remain in the study until after delivery and discharge from hospital for the mother and baby, or 1 month after delivery, whichever comes first. Outcomes will be collected from electronic records.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Being induced
* Singleton pregnancy
* Primiparous
* ≥37+0 weeks gestation
* Intact membranes
* Able to provide informed consent

Exclusion criteria:

* Previous cervical surgery
* Any cervical pathology at 12 o'clock position on cervix
* Vaginal bleeding evident on examination
* Visible, symptomatic cervical or vaginal infections
* Known congenital uterine anomalies
* Known or suspected structural/chromosomal fetal abnormality
* Known HIV
* Cervical carcinoma

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female of reproductive age with confirmed singleton pregnancy.
Study Population: Participants with singleton, term pregnancy, requiring induction of labour.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with Vaginal Delivery | 5 days (time of commencing induction of labour to outcome of delivery)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sharp, Study Director — University of Liverpool
Locations (1):
- Liverpool Women's Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medford E, Lane S, Merriel A, Sharp A, Care A. The CASPAR study protocol. Can cervical stiffness predict successful vaginal delivery after induction of labour? a feasibility, cohort study. PLoS One. 2025 Jan 16;20(1):e0311324. doi: 10.1371/journal.pone.0311324. eCollection 2025. PMID 39820788
- See also: Cervical stiffness assessment device website Available IPD/Information: — http://en.pregnolia.com/